CLINICAL TRIAL: NCT03911466
Title: NIDA CTN Protocol 0080: Medication Treatment for Opioid Use Disorder in Expectant Mothers (MOMs): a Pragmatic Randomized Trial Comparing Extended-release and Daily Buprenorphine Formulations: Conceptual Model Assessments (CMA) Sub-study
Brief Title: Medication Treatment for Opioid Use Disorder in Expectant Mothers: Conceptual Model Assessments Sub-study
Acronym: MOMs-CMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: T. John Winhusen, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, T. John Winhusen, PhD, Professor; Vice Chair and Division Director of Addiction Sciences, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0429-2; UG1DA013732 (NIH)
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Opioid-Related Disorders; Drug Addiction; Pregnancy Related; Substance Abuse; Drug Abuse; Neonatal Abstinence Syndrome; Neonatal Opioid Withdrawal Syndrome; Drug Abuse in Pregnancy
Keywords: CTN-0080; clinical trials network; medication assisted treatment; pharmacokinetics
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Neonatal Abstinence Syndrome | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BUP-XR (Experimental): Weekly subcutaneous Buprenorphine Injection (CAM2038) during pregnancy. During the 12-month postpartum phase, participants who are breastfeeding will continue receiving subcutaneous Buprenorphine Injection weekly; participants who are not breastfeeding will receive subcutaneous Buprenorphine Injection monthly.
  The target doses will be 24 mg for the weekly formulation and 96 mg for the monthly formulation, but the actual dose may be lower or higher as determined by the prescribing clinician (e.g., based on craving/withdrawal experienced by the participant, etc.).
  Interventions: Drug: Buprenorphine Injection
- BUP-SL (Active Comparator): Daily sublingual buprenorphine, with or without naloxone, based on site preference, during pregnancy and during the 12-month postpartum phase.
  The target dose will be 16 mg daily, but the actual dose may be lower or higher as determined by the prescribing clinician (e.g., based on craving/withdrawal experienced by the participant, etc.).
  Interventions: Drug: Buprenorphine Sublingual Product

INTERVENTIONS:
Drug: Buprenorphine Injection — Weekly and monthly formulations of injectable, extended-release buprenorphine (BUP-XR).
  Other Names: CAM2038
  Arms: BUP-XR
Drug: Buprenorphine Sublingual Product — Sublingual buprenorphine (BUP-SL), administered daily.
  Other Names: Subutex; Suboxone
  Arms: BUP-SL

SUMMARY:
This is a sub-study of NIDA CTN Protocol 0080: Medication Treatment for Opioid Use Disorder in Expectant Mothers (MOMs; Unique protocol ID: 2019-0429-1). Participants in MOMs will be offered the opportunity to enroll in this sub-study, which is designed to evaluate conceptual models of the mechanisms by which extended-release buprenorphine (BUP-XR), may improve mother-infant outcomes, compared to sublingual buprenorphine (BUP-SL). The additional data collected in this sub-study will be combined with data from the main MOMs trial.

It is hypothesized that: (1) the buprenorphine blood levels will vary, depending on which formulation of buprenorphine was received, (2) the variation in buprenorphine blood levels will be associated with fetal behavior (including fetal heart rate variability) (3) the variation in buprenorphine blood levels will be associated with differences in mother outcomes (including medication adherence and illicit opioid use) (4) the variation in buprenorphine blood levels and in fetal behavior will be associated with infant outcomes (including neonatal opioid withdrawal syndrome and infant development).

ELIGIBILITY:
Inclusion Criteria:

* Participating in the MOMs trial (Unique protocol ID: 2019-0429-1)

Exclusion Criteria:

-

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Cmin of buprenorphine and metabolites in plasma | 2 weeks post-randomization
  A blood draw at the estimated time of minimum drug concentration ("trough") to evaluate adequacy of dose for the conceptual model.
Cmin of buprenorphine and metabolites in plasma | 4 weeks post-randomization
  A blood draw at the estimated time of minimum drug concentration ("trough") to evaluate adequacy of dose for the conceptual model.
Fetal heart rate variability | Estimated gestational age (EGA) approximately 36 weeks
  This is the measure of primary interest from the fetal evaluation (non-stress test and biophysical profile).
Cmin of buprenorphine and metabolites in plasma | Estimated gestational age (EGA) approximately 36 weeks
  A blood draw at the estimated time of minimum drug concentration ("trough") to evaluate trough-to-peak fluctuation for the conceptual model.
Cmax of buprenorphine and metabolites in plasma | Estimated gestational age (EGA) approximately 36 weeks
  A blood draw at the estimated time of maximum drug concentration ("peak") to evaluate trough-to-peak fluctuation for the conceptual model.
Concentration of buprenorphine and metabolites in maternal plasma | Delivery
  A blood draw around the time of delivery to evaluate the association between drug concentration and neonatal opioid withdrawal syndrome outcomes.
Concentration of buprenorphine and metabolites in cord plasma | Delivery
  Cord blood will be collected and used to estimate fetal exposure to buprenorphine.

CONTACTS AND LOCATIONS:
Overall Officials: T. John Winhusen, PhD, Principal Investigator — University of Cincinnati
Locations (12):
- United States (12):
  - Gateway Community Services, Jacksonville, Florida
  - Massachusetts General Hospital HOPE Clinic, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of New Mexico Milagro Clinic, Albuquerque, New Mexico
  - University of Cincinnati Health Perinatal Addictions Program, Cincinnati, Ohio
  - CODA, Inc., Portland, Oregon
  - Pregnancy Recovery Center at Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah SUPeRAD Clinic, Salt Lake City, Utah
  - Addiction Recovery Services (ARS), Swedish Medical Center, Seattle, Washington
  - Marshall Health MARC Program, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data will be transmitted by the study Data and Statistics Center to the designated party for de-identification, posting, storing, and archiving on NIDA's Data Share website. Data Share is an online repository of data from studies funded by the National Institute on Drug Abuse. All de-identified individual participant data is expected to be made available.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Kropp FB, Smid MC, Lofwall MR, Wachman EM, Martin PR, Murphy SM, Wilder CM, Winhusen TJ. Collaborative care programs for pregnant and postpartum individuals with opioid use disorder: Organizational characteristics of sites participating in the NIDA CTN0080 MOMs study. J Subst Use Addict Treat. 2023 Jun;149:209030. doi: 10.1016/j.josat.2023.209030. Epub 2023 Apr 4. PMID 37023858

DOCUMENTS (1):
  • Informed Consent Form (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT03911466/ICF_001.pdf